CLINICAL TRIAL: NCT02387060
Title: Use of Intrathecal Fentanyl and Development of Hyperalgesia in Patients Undergoing Elective Cesarean
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-389
Record Dates: First submitted 2015-02-25; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Complications; Cesarean Section
Keywords: Anesthesia; Spinal and Epidural; Adverse Effect; Complications
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- H-Bupivacaine 11.5 mg + fentanyl 25 mcg. (Experimental): Intrathecal administration of Hyperbaric Bupivacaine 1.5 ml 0.75% plus fentanyl 25 mcg.
  Interventions: Drug: H-Bupivacaine; Drug: Fentanyl
- H-Bupivacaine 11.5 mg. (Active Comparator): Intrathecal administration of Hyperbaric Bupivacaine 1.5 ml 0.75%
  Interventions: Drug: H-Bupivacaine

INTERVENTIONS:
Drug: H-Bupivacaine — Intrathecal administration of hyperbaric bupivacaine 1.5 ml 0.75%
  Other Names: Hyperbaric bupivacaine
Drug: Fentanyl — Intrathecal administration of fentanyl 25 mcg
  Arms: H-Bupivacaine 11.5 mg + fentanyl 25 mcg.

SUMMARY:
Opioid analgesic drugs are the main treatment of patients during anesthesia. Although highly effective, their use is not without problems. One is the increasing requirement of these address the same nociceptive stimulus.

Opioid induced hyperalgesia could be an explanation studies in animal models. Through mechanisms where N-methyl-D-aspartate receptors, glutamatergic system disturbances and changes in intracellular calcium regulation involved.

The hyperalgesia induced by intrathecal opioids is controversial. The investigators propose a model study in patients undergoing cesarean section to study the secondary hyperalgesia induced based on the study of nociceptive thresholds with two methods opioids: Von Frey filaments and digital algometer.

If intrathecal fentanyl is used in spinal anesthesia for elective cesarean section, then, an increase in sensitivity will occur. This increase can be measured by von Frey filaments, expressed in increased requirement clinically opioids.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant 37 to 41 weeks.
* American Society of Anesthesiologists classificationI or II.
* Between 18 and 40 years.
* Scheduled for elective cesarean section under spinal anesthesia in the Maternity Service of the Clinical Hospital of the Catholic University.

Exclusion Criteria:

* Background Of high risk pregnancy. Twin-pregnancy.
* Obesity> 30 kg / m 2 before pregnancy.
* Background Of psychiatric illness.
* Using Chronic analgesic.
* AllergyDrug used in protocol.
* require General anesthesia during surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in Punctate - Von frey (grams) | Change from Baseline in punctate sensibility at 48 hours

SECONDARY OUTCOMES:
Change in Pressure pain - algometer (kg/cm/cm) | Change from Baseline in pressure pain at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortinez, MD, Study Chair — Ponticia Universidad Católica
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica, Santiago, Santiago Metropolitan, Chile